CLINICAL TRIAL: NCT06692595
Title: Digital PCR for Quantifying Periodontal Pathobionts: A Comparative Study With qPCR
Brief Title: Digital PCR for Quantifying Periodontal Pathobionts
Acronym: dPCR
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Rok Gašperšič, Assoc. Prof., PhD, University of Ljubljana
Other Study IDs: UKCdPCR1; J7-4639 (Other Grant/Funding Number: ARIS)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Subgingival plaque sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis patients
  Interventions: Diagnostic Test: digital PCR
- Individuals with healthy periodontium
  Interventions: Diagnostic Test: digital PCR

INTERVENTIONS:
Diagnostic Test: digital PCR — digital PCR quantification of subgingival plaque samples

SUMMARY:
Comparison of quantitative polymerase chain reaction (qPCR) and digital polimerase chain reaction (dPCR) quantification of subgingival plaque samples.

ELIGIBILITY:
For inclusion, each subject had to be systemically healthy and aged 20 to 80 years. Subjects were excluded if they: had less than 5 teeth in each jaw quadrant, regularly used a mouthwash as part of their oral hygiene routine, had received antibiotics during the last 6 months or during the study period, were pregnant or lactating, had a known systemic illness (i.e. HIV/AIDS, diabetes mellitus, cancer, diseases of bone metabolism, diseases affecting wound healing) or were treated with immunosuppressants, chemotherapy, radiation, calcium antagonists, antiepileptics and non-steroidal anti-inflammatory drugs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study comprised of two subject groups. The first group consisted of 20 subjects with periodontitis, who had at least one probing site in each jaw quadrant with pocket depth (PPD) measuring > 4 mm and positive bleeding on probing (BOP). Periodontitis stage and grade were determined following the 2018 classification system.
  The second group consisted of 20 volunteers without periodontal pathologies (healthy group), i.e. plaque index < 10% at baseline visit, absence of periodontal pockets measuring > 4 mm and no prior periodontal treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
concentration of targeted bacterial species, expressed as genome equivalents per mL (Geq/mL), normalized for ribosomal gene copy number per cell | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No